CLINICAL TRIAL: NCT01942980
Title: Double-blind Randomized Multicenter Phase III Study Evaluation of the Efficacy of Hippocampal Avoidance on the Cognitive Toxicity of Whole-brain Radiation Therapy After Surgical Resection of Single Brain Metastasis of Breast Cancer.
Brief Title: Evaluation of the Efficacy of Hippocampal Avoidance on the Cognitive Toxicity of Whole-Brain Radiation Therapy After Surgical Resection of Single Brain Metastasis of Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHIToN / IPC 2012-005
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Brain Metastasis
Keywords: Breast cancer; one brain metastasis
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional postoperative whole-brain radiation therapy (Other): conventional postoperative whole-brain radiation therapy (40 Gy in 20 fractions of 2 Gy)
  Interventions: Radiation: Radiation therapy Brain metastasis in breast cancer
- whole-brain radiation therapy with hippocampal avoidance (Other): Radiation therapy with hippocampal avoidance
  Interventions: Radiation: Radiation therapy Brain metastasis in breast cancer

INTERVENTIONS:
Radiation: Radiation therapy Brain metastasis in breast cancer — Radiation

SUMMARY:
The incidence of brain metastases (BM) in metastatic breast cancer is increasing, due to the improvement in the control of systemic disease, and due to an improved detection through imagery.

The treatment management of single BM remains controversial. Indeed, even though it is widely accepted that local treatment increases the median survival time in patients having a good prognostic status, the adding of "adjuvant" whole-brain radiation therapy (WBRT) is currently subject to controversy, due to its potential toxicity. Yet, two randomized trials have demonstrated a clear increase in intra-cerebral recurrence and in death from neurologic origin in case of absence of "adjuvant" WBRT, without change in overall survival (but overall survival was not a primary endpoint in any of these studies).

The data from literature on cognitive toxicity (CT) of WBRT on BM are scarce and sometimes controversial. CT of WBRT affects the subcortical frontal functions. It is postulated that the alteration of hippocampal neurogenesis (mainly due to inflammation process), situated in the subgranular zone of the dentate gyrus, has an essential role in the development of these brain dysfunctions.

It has been shown that the incidence of BM in the hippocampal region (hippocampus + 5mm expansion) is low, in the range of 8,6%.

New irradiation techniques, in particular intensity-modulated radiotherapy associated with rotational radiotherapy, allow to modulate the dose on an intra-cerebral structure, all the while distributing an adapted dose to the remaining brain.

This prospective, randomized study, will compare, through a battery of neuropsychological tests, the cognitive impact of WBRT of 40 Gy in 20 fractions with or without hippocampal avoidance by intensity modulated radiotherapy, in patients presenting with a single operated brain metastasis of breast cancer. If the hippocampal avoidance leads to a significant improvement in cognitive function, this radiotherapy scheme could become the standard postoperative treatment to be proposed to patients presenting the best prognostic factors. This would allow to prevent long-term cognitive deficit, while preserving WBRT benefit on intra-cerebral control.

Justification of evaluation criteria :

Principal criteria :

Evaluation criteria to assess cognitive toxicity have been selected on the basis of the recommendations from C. Meyers and P. Brown, who propose an adapted test battery to evaluate memory, verbal function, visual and motor coordination, and executive function. The selected tests have been validated, also in French. They comprise HVLT-R (Hopkins Verbal Learning Test Revised), COWAT (Controlled Oral Word Association Test), Grooved Pegboard test, TMT A and B (Trailmaking tests A and B), and MMSE. The calculation of patient numbers was based on the HVLT-R test, as memory is thought to be the most frequently affected domain.

The tests will be performed before treatment ("baseline" cognitive function), at 4 months and at 12 months. In case of a missing answer to the evaluation tests, the reason(s) for not answering will be noted.

Secondary criteria :

Quality of life : QLQ-C30, QLQ-BN20, ADL, IADL Intra-cerebral Progression-free survival (PFS) Overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal 18 years old,
* Single brain metastasis from breast cancer, first cerebral event,
* Complete surgical resection of cerebral metastasis,
* Histological confirmation of brain metastasis of breast cancer,
* Start of radiotherapy within 6 weeks after surgery,
* Karnofsky > or equal to 70,
* No history of brain radiotherapy,
* Signed informed consent to participate,
* Patient affiliated to a social security system or benefiting from such a system.

Exclusion Criteria:

* Multiple brain metastases, leptomeningeal metastases,
* macroscopic metastasis surgery not complete,
* Warning signs of brain displacement (uncontrolled oedema),
* History of cerebral irradiation or absence of surgical treatment of the current metastasis,
* History of cancer in the previous 5 years prior to entry in the study, other than cutaneous basal cell carcinoma or in situ epithelioma of uterine cervix or the stated breast cancer,
* MMSE (Mini Mental State Examination)< 24,
* all previous systemic treatments less than 2 weeks are not allowed,
* Pregnant women or liable to become pregnant, lactating women,
* Persons deprived of their freedom or under tutelage
* Patients unable to comply with medical procedures of the study for geographical, social, or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03-22 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
To assess cognitive toxicity | From inclusion/randomization to 12 months
  Evaluation criteria to assess cognitive toxicity have been selected on the basis of the recommendations from C. Meyers and P. Brown, who propose an adapted test battery to evaluate memory, verbal function, visual and motor coordination, and executive function. The selected tests have been validated, also in French. They comprise HVLT-R (Hopkins Verbal Learning Test Revised), COWAT (Controlled Oral Word Association Test), Grooved Pegboard test, TMT A and B (Trailmaking tests A and B), and MMSE. The calculation of patient numbers was based on the HVLT-R test, as memory is thought to be the most frequently affected domain.

SECONDARY OUTCOMES:
Quality of life | At inclusion/randomization, at month 1, month 4 and month 12
  Quality of life : QLQ-C30, QLQ-BN20, ADL, IADL. Intra-cerebral Progression-free survival (PFS) up to 24 months. Overall survival up to 24 months.
Intra-cerebral progression | Evaluated every 3 months
  to assess by RMI or clinical signs
Overall survival | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Agnès TALLET, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Agnès TALLET, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr